CLINICAL TRIAL: NCT01265992
Title: Post Marketing Observational Study to Assess Patient Management Practices and Quality of Life With the Capsules Form of Paricalcitol in the Treatment of SHPT in Stage 3 - 5 Chronic Kidney Disease Patients Not Yet on Dialysis Under Conditions of Usual Clinical Care (CAPITOL)
Brief Title: Study to Assess Patient Management Practices and Quality of Life With Paricalcitol Capsules in the Treatment of Secondary Hyperparathyroidism in Stage 3-5 Chronic Kidney Disease Patients Not Yet on Dialysis
Acronym: CAPITOL
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-270
Record Dates: First submitted 2010-11-29; First posted 2010-12-24 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-01

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: Secondary hyperparathyroidism; Mineral and Bone Disorder (CKD-MBD); Chronic Kidney Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Calcinosis; Bone Diseases; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paricalcitol capsules: Patients with secondary hyperparathyroidism associated with Stage 3 - 5 CKD and not yet on dialysis and prescribed paricalcitol capsules in accordance with the terms of the marketing authorization in Sweden.

SUMMARY:
Paricalcitol capsules (Zemplar®) received marketing authorization in Sweden in late 2007 for the prevention and treatment of secondary hyperparathyroidism in patients with Stage 3 & 4 Chronic Kidney Disease (CKD). Accordingly, additional data is needed to evaluate the effectiveness and safety of paricalcitol therapy under conditions of usual clinical care in Sweden.

This observational study is designed to collect data to evaluate safety and effectiveness during 6 months of therapy with paricalcitol capsules prescribed for patients with CKD Stages 3-5 not yet on dialysis. Data will also be collected on patient quality of life and costs associated with patient care.

DETAILED DESCRIPTION:
This observational study is designed to collect data to evaluate safety and effectiveness during 6 months of therapy with paricalcitol capsules prescribed in accordance with the terms of the marketing authorization for patients with Chronic Kidney Disease (CKD) Stages 3-5 not yet on dialysis. Data will also be collected on patient quality of life and costs associated with patient care. A retrospective chart review of patient laboratory and medication history will provide historical data to determine drivers for initiation of paricalcitol therapy.

The primary goal of this post-marketing observational study (PMOS) is to further characterize the prescribing habits and patient management practices of physicians prescribing paricalcitol capsules and to assess the metabolic safety and effectiveness of paricalcitol capsules for the treatment of secondary hyperparathyroidism in Stage 3-5 CKD patients not yet on dialysis under conditions of usual clinical care. Focus will be to examine the practice of dose titration in early stages of CKD, understand real-world management of intact parathyroid hormone levels, understand real-world incidence and management of abnormalities in serum calcium and phosphate, and to examine patient bone and mineral profiles and medical history to understand drivers for paricalcitol capsules use.

Patients prescribed paricalcitol therapy for the first time will be asked to participate in the study. Enrolled patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

Patients must sign the Informed Consent Form prior to inclusion into the study

* Patients should satisfy the Swedish Summary of Product Characteristics (SPC) for paricalcitol capsules at www.fass.se
* Patients must be 18 years or older with a diagnosis of secondary hyperparathyroidism associated with Chronic Kidney Disease (CKD) Stages 3 - 5 (estimated Glomerular Filtration Rate between 10-59 by Modification of Diet in Renal Disease) but not yet on dialysis
* Patients should be in stable condition and have a life expectancy of at least 6 months
* Patients should not be expected to be transplanted or initiate dialysis for at least 6 months

Exclusion Criteria:

* Patients with CKD receiving dialysis
* Patients contraindicated for paricalcitol capsules as described in the SPC
* Treatment with paricalcitol more than 20 days prior to study enrollment
* History of drug or alcohol abuse within 6 months prior to inclusion
* History of non-compliance with medication or a medical history (i.e. psychiatric) that could enhance non-compliance with medication as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals with nephrology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Dahl, MD, Study Director — AbbVie
Locations (10):
- Sweden (10):
  - Site Reference ID/Investigator# 47723, Kalmar
  - Site Reference ID/Investigator# 41084, Karlstad
  - Site Reference ID/Investigator# 45190, Kristianstad
  - Site Reference ID/Investigator# 41085, Linköping
  - Site Reference ID/Investigator# 41087, Norrköping
  - Site Reference ID/Investigator# 45188, Örebro
  - Site Reference ID/Investigator# 41088, Skövde
  - Site Reference ID/Investigator# 57782, Stockholm
  - Site Reference ID/Investigator# 41089, Värnamo
  - Site Reference ID/Investigator# 45191, Västerås

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Paricalcitol Capsules: Patients with secondary hyperparathyroidism associated with Stage 3 - 5 chronic kidney disease (CKD) and not yet on dialysis and prescribed paricalcitol capsules in accordance with the terms of the marketing authorization in Sweden.
Period: Overall Study
Arm/Group | Paricalcitol Capsules
Started | 50
Received Treatment | 49
Completed | 41
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Administrative reasons | 2
Not completed — Stopped treatment | 3
Not completed — Did not receive treatment | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set, defined as all included participants who received at least 1 dose of paricalcitol capsules.
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  White | 49
  Black | 0
  Asian | 0
  American (Indian/Alaska Native) | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 49

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intact Parathyroid Hormone at 6 Months
Time Frame: Baseline and 6 months
Population: Per-Protocol Analysis Set (PPAS), defined as all included participants who received at least 1 dose of paricalcitol capsules and had analyzable data for the primary endpoints, i.e., 5 - 8 months after inclusion, and with available iPTH data at both time points.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 36
pmol/L | -6.2 (13.0)

2. Primary Outcome: Percentage of Participants With Intact Parathyroid Hormone Within K/DOQI Target Range at Baseline and 6 Months
Description: Kidney Disease Outcomes Quality Initiative (K/DOQI) target intact parathyroid hormone (iPTH) levels are:
  Stage 3 CKD (estimated Glomerular Filtration Rate* [eGFR] 30 - 59 mL/min): 3.85 - 7.7 pmol/L;
  Stage 4 CKD (eGFR 15 - 29 mL/min): 7.7 - 12.1 pmol/L;
  Stage 5 CKD (eGFR < 15 mL/min): 16.5 - 33 pmol/L.
  *Calculated using the Modification of Diet in Renal Disease formula.
Time Frame: Baseline and 6 months
Population: Per-protocol analysis set. Three participants had missing data at Baseline and one participant had missing data at the 6 month visit; percentages are based on the total number of participants in the per-protocol analysis set (40).
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 40
percentage of participants
  Baseline | 15.0
  6 months | 27.5

3. Primary Outcome: Percentage of Participants With Elevated Serum-Phosphorus (s-P) Levels at Baseline and 6 Months
Description: Elevated serum phosphorus is defined according to the 2003 Kidney Disease Outcomes Quality Initiative (K/DOQI) target definitions as:
  Stage 3 CKD: ≥ 1.49 mmol/L;
  Stage 4 CKD: ≥ 1.49 mmol/L;
  Stage 5 CKD: > 1.78 mmol/L.
Time Frame: Baseline and 6 months
Population: Per-protocol analysis set. Two patients had missing s-P data at month 6; percentages are based on the total number of participants in the per-protocol analysis set (40).
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 40
percentage of participants
  Baseline | 15.0
  6 months | 25.0

4. Primary Outcome: Percentage of Participants With Elevated Serum-Calcium (s-Ca) Levels at Baseline and 6 Months
Description: Elevated serum calcium is defined according to the 2003 Kidney Disease Outcomes Quality Initiative (K/DOQI) target definitions of s-Ca above 2.37 mmol/L.
Time Frame: Baseline and 6 months
Population: Per-protocol analysis set. One participant had missing s-Ca data at Baseline and one participant had missing s-Ca data at month 6; percentages are based on the total number of participants in the per-protocol analysis set (40).
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 40
percentage of participants
  Baseline | 42.5
  6 months | 42.5

5. Secondary Outcome: Change From Baseline in Proteinuria
Description: Proteinuria is the presence of excess serum proteins, or albumin, in the urine. Proteinuria was measured by the amount of albumin per liter of urine.
Time Frame: Baseline and Month 6
Population: Per-protocol analysis set with available data at both time points.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 10
g/L | 0.2 (0.7)

6. Secondary Outcome: Percentage of Participants With a Reduction of Proteinuria of at Least 15% From Baseline
Time Frame: Baseline and 6 months
Population: Per-protocol analysis set. Percentages are based on the total number of participants in the per-protocol analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 40
percentage of participants | 10.0

7. Secondary Outcome: Change From Baseline in Quality of Life Assessed by the Kidney Disease Quality of Life-Short Form (KDQOL-SF)
Description: The KDQOL-SF is a self-report measure developed for individuals with kidney disease. It includes 43 end-stage renal disease (ESRD)-targeted items focused on particular areas of concern for individuals with kidney disease (Symptoms/problems, Effects of the disease on daily life, Burden of disease, Work status, Cognitive function, Quality of social interaction, Sexual function, Sleep, and Social support), 36 items (SF-36) that provide 8 measures of physical and mental health (Physical functioning, Role limitations caused by physical health limitations, Role limitations caused by emotional health problems, Social functioning, Emotional well-being, Pain, Energy/fatigue and General health perceptions), and 1 overall health rating item where respondents rate their health on a scale from 0 ("worst possible health") to 10 ("best possible health").
  Scores are transformed and calculated such that each scale score ranges from 0 to 100 where higher scores reflect a better quality of life.
Time Frame: Baseline and 6 months
Population: Per-protocol analysis set with available data at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 24
units on a scale
  ESRD: Symptom/problem scale | -0.4 (12.9)
  ESRD: Effects of kidney disease | -0.2 (9.4)
  ESRD: Burden of kidney disease | -1.0 (19.5)
  ESRD: Work status | -10.4 (29.4)
  ESRD: Cognitive function | -2.5 (19.7)
  ESRD: Quality of social interaction | 1.7 (20.3)
  ESRD: Sexual function | -0.6 (23.0)
  ESRD: Sleep | 0.9 (11.3)
  ESRD: Social Support | -4.9 (17.4)
  SF-36: Physical functioning | 5.7 (18.6)
  SF-36: Role physical | -7.3 (36.5)
  SF-36: Pain | -2.3 (22.1)
  SF-36: General health | 1.5 (16.6)
  SF-36: Emotional well-being | -3.0 (13.4)
  SF-36: Role emotional | -11.1 (36.3)
  SF-36: Social function | 0.5 (22.0)
  SF-36: Energy/fatigue | 1.9 (22.4)
  Overall health rating | 1.3 (15.4)

8. Secondary Outcome: Total Direct Costs of Care Associated With Secondary Hyperparathyroidism
Description: Direct medical costs to be calculated included outpatient visits, hospitalizations, pharmaceuticals, etc. However the data collected in this observational study was not enough to support this calculation.
Time Frame: 6 months
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 0

9. Secondary Outcome: Total Indirect Costs of Care Associated With Secondary Hyperparathyroidism
Description: Indirect costs were estimated by using the number of hours missed from work (absenteeism) multiplied by the average hourly labor cost, including wages and benefits, to calculate average lost productivity costs due to absenteeism during the preceding 7 days.
  Hours missed from work were assessed using the Work Productivity and Activity Impairment Questionnaire: General Health (WPAI-GH) questionnaire, in which respondents answer 6 questions related to work productivity and impairment.
  Unit costs were taken from official sources (Statistics Sweden, www.scb.se) and published literature.
Time Frame: 6 months
Population: Participants who were working for pay and with available data at both time points.
Measure: Mean (Standard Deviation); unit: Swedish krona per participant
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 11
Swedish krona per participant
  Absenteeism: Baseline | 0 (0)
  Absenteeism: 6 months | 1,318 (2,642)

10. Secondary Outcome: Number of Participants Using Concomitant Medications at Baseline
Time Frame: Baseline
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Paricalcitol Capsules
Number analyzed (Participants) | 49
participants
  Agents acting on the renin-angiotensin system | 39
  All other therapeutic products | 11
  Angiotensin II antagonists, plain | 1
  Antianemic preparations | 10
  Antigout preparations | 9
  Antihypertensives | 5
  Antiprotozoals | 1
  Antithrombotic agents | 2
  Beta blocking agents | 22
  Blood substitutes and perfusion solutions | 10
  Calcium channel blockers | 27
  Calcium homeostasis | 1
  Cardiac therapy | 1
  Diuretics | 28
  Drugs for obstructive airway diseases | 1
  Drugs used in diabetes | 3
  Immunosuppressive agents | 1
  Lipid modifying agents | 28
  Mineral supplements | 10
  Vitamins | 2

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only Serious Adverse Events (SAEs) were collected in this Post Marketing Observational Study.
Arm/Group | Paricalcitol Capsules
Serious Adverse Events (participants affected / at risk) | 12/49
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Capsules (N=49)
Acute myocardial infarction (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 2
General physical health deterioration (General disorders) | 2
Pyrexia (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Ageusia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Coordination abnormal (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Anuria (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Aortic aneurysm rupture (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Poor peripheral circulation (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.